CLINICAL TRIAL: NCT03505424
Title: Supporting All Families of Premature Infants At Prentice Women's Hospital from Admission Through Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Friends of Prentice (Other)
Responsible Party: Principal Investigator, Craig Garfield, Associate Professor in Pediatrics, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00207127
Record Dates: First submitted 2018-03-30; First posted 2018-04-23 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Premature Infant; Premature Birth; NICU
Keywords: Premature Infant; Premature Birth; Smartphone App; NICU
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Standard of Care (Active Comparator): Parents of infants born from April -mid-August 2018 (Group 1)
  Interventions: Other: Group 1: Standard of Care
- Group 2: NICU2HOME app (Active Comparator): Parents of infants born from mid-August 2018- January 2019 (Group 2)
  Interventions: Other: Group 2: NICU2HOME app
- Group 3: SMART NICU2HOME app (Active Comparator): Parents of infants born from February- June 2019 (Group 3)
  Interventions: Other: Group 3: SMART NICU2HOME app

INTERVENTIONS:
Other: Group 1: Standard of Care — Those who are in Group 1 will receive the usual care which includes:
  1. a welcome packet from the nursing staff
  2. access to their infant's medical team including doctors and nurse
  3. opportunities to ask any questions and understand the care their baby is receiving through participation in daily work rounds or through setting up family meetings with the medical team.
  Arms: Group 1: Standard of Care
Other: Group 2: NICU2HOME app — In addition to the usual care made available to Group 1 as described above, Group 2 parents will receive the smartphone app. Group 2 parents will be asked to download the NICU2HOME app.
  Arms: Group 2: NICU2HOME app
Other: Group 3: SMART NICU2HOME app — In addition to the usual care made available to Group 1 as described above, Group 2 parents will receive the smartphone app. Group 3 parents will be asked to download the SMART NICU2HOME app.
  Arms: Group 3: SMART NICU2HOME app

SUMMARY:
The objective of this study is to determine the extent to which the SMART NICU2HOME (including EMR interface) and the NICU2HOME apps, mobile applications designed for parents of premature infants to receive daily, real-time information about their infants and personalized education material based on parents' anticipated concerns and their infant's clinical status, is effective in: 1) improving parents' competency in caring for their sick infants, 2) reducing stress, 3) supporting parents' social supports and 3) improving NICU outcomes (parent satisfaction, length of stay, readmission rates.)

DETAILED DESCRIPTION:
There will be four groups of participants based on when the infant is in the NICU.

Parents of infants born from April -Mid-August 2018 (Group 1) Group 1 participants will receive usual care which includes 1) a welcome packet from the nursing staff, 2) access to their infant's medical team including doctors and nurse, 3) opportunities to ask any questions and understand the care their baby is receiving through participation in daily work rounds or through setting up family meetings with the medical team.

At NICU admission, parents in Group 1 will be asked to complete a brief demographics form and several standardized surveys that measure stress and life experiences. Surveys will again be administered 7-10 days later, the day before discharge, two weeks after discharge and 30 days after discharge. These surveys will be available both via on paper or an email link.

Parents of infants born from Mid-August - January 2019 (Group 2) At NICU admission, parents in Group 2 will be asked to complete a brief demographics form and several standardized surveys that measure stress and life experiences. Surveys will again be administered 7-10 days later, the day before discharge, two weeks after discharge and 30 days after discharge. These surveys will be available both via on paper or an email link.

In addition to the usual care made available to Group 1 and described above, Group 2 parents will also be asked to download the NICU2HOME app from a given website where they will enter MRN, DOB, name, gender, and due date of their infant into the smartphone app. In case there are difficulties downloading or using the app, the research team will be available to assist parents with any questions or concerns.

Parent of infants born from February 2019- June 2019 (Group 3) At NICU admission, parents in Group 3 will be asked to complete a brief demographics form and several standardized surveys that measure stress and life experiences. Surveys will again be administered 7-10 days later, the day before discharge, two weeks after discharge and 30 days after discharge. These surveys will be available both via on paper or an email link. In addition to the usual care made available to Group 1, Group 3 parents will also be asked to download the SMART NICU2HOME app from a given website where they will enter MRN, DOB, name, gender, and due date of their infant into the smartphone app.

Parent of infants born from November 2019- December 2020 (Group 4) At NICU admission, parents in Group 4 will be asked to complete a brief demographics form and several standardized surveys that measure stress and life experiences as well as parental efficacy. Surveys will again be administered 30 and 60 days later depending on the gestational age of the baby, the day of discharge, two weeks after discharge and 30 days after discharge. These surveys will be available through an email link.

In addition to the usual care made available to Group 1 and described above, Group 4 parents will also be asked to download the NICU2HOME app from a given website where they will enter MRN, DOB, name, gender, and due date of their infant into the smartphone app. In case there are difficulties downloading or using the app, the research team will be available to assist parents with any questions or concerns. Participants in Group 4 will not be paid for their contribution to the research.

Each participant (in both groups) will be asked to complete the surveys independently without sharing responses. If completed on paper, the research team will arrange either to pick the survey up at the NICU if the baby is still in the hospital, via a pre-paid stamped envelope provided, or over the phone. Online surveys will be automatically returned.

Optional Interview:

In addition to the intervention study, an optional qualitative interviews will be conducted with 30 families from group 2 and group 3 for about 30-45 minutes. Patients will have the option to opt to participate in the interviews when consenting to the main study by signing their initials on the "Optional Elements" to be interviewed. Consenting to be interviewed also means that they have agreed to let us audio record the interview for research purposes. Of those who opted to be interviewed, only 30 families will be randomly selected to partake in the interviews.

Using maximum variation sampling method, the interview will occur around 1-2 days prior to discharge (final thoughts, use patterns) with approximately 5 families per gestational age bracket: <28 weeks; 28-<30 weeks; 30-<32 weeks; 32-<34 weeks; 34-<37 weeks. The interviews will be semi-structured, one-on-one phone on in-person interviews (option is the family's) designed to elicit feature feedback reasons for their level of usage. With consent, all interviews will be audio-recorded, transcribed, coded, and analyzed for themes to improve further iterations. These audio recordings (either in voice or transcription) may be used in scholarly presentations or publications serve to help other professionals understand the research. No identifiers will be present when sharing the recordings to maintain anonymity, and recordings will be saved with a study ID number rather than name.

NICU2HOME app was created for parents of premature infants to meet their demands. The app will teach parents about their baby and the NICU. It will allow them to receive educational material every day that is specifically geared towards their baby's journey in the NICU. The app will also all parents to connect with their friends and family allowing them to privately and safely share and post among themselves.

SMART NICU2HOME app includes the same features and functions as the NICU2HOME app stated above; however, it also allows parents to receive a daily update of the clinically benign information of their infant directly from the EPIC EMR, such as, days of life, adjusted gestational age, weight, length, etc.

ELIGIBILITY:
Inclusion Criteria:

* Parents of premature infants (<37 weeks) admitted to Prentice NICU
* Competent in English (i.e. to fully understand the questions asked in the surveys)
* Smartphone owner

Exclusion Criteria:

* None Adults unable to consent/Cognitively Impaired
* Pregnant women (where the activities of the research may affect the pregnancy or the fetus)
* Prisoners or other detained individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the level of confidence caring for their premature infants while in the NICU and once at home measured through a survey. | 2-3 months
  We will use the PSOC Survey for this outcome.

SECONDARY OUTCOMES:
The primary outcome measure will be the level of stress caring for their premature infants while in the NICU and once at home measured through a survey. | 2-3 months
  We will use the PSS Survey for this outcome.
Relationship quality will be measured through survey. | 2-3 months
  We will use the MOS Survey for this outcome.

OTHER OUTCOMES:
Patient satisfaction with the hospitalization will be measured through survey. | 2-3 months
  We will use the Press Gainey Survey for this outcome.
Patient satisfaction with the discharge will be measured through survey. | 2-3 months
  We will use the Press Gainey Survey for this outcome.
Social support will be measured through survey. | 2-3 months
  We will use the MOS Survey for this outcome.
Length of Stay will be measure. | 2-3 months
  We will calculate the length of stay in the hospital on the admission and discharge collection sheets.
Readmission rates will be measure. | 2-3 months
  We will gather this information in our post discharge survey,

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamilton BE Ph D, Martin JA, Osterman MJ M H S, Curtain SC M A. Births: Preliminary Data for 2014. Natl Vital Stat Rep. 2015 Jun;64(6):1-19. PMID 26114874
- [Background] Institute of Medicine (US) Committee on Understanding Premature Birth and Assuring Healthy Outcomes; Behrman RE, Butler AS, editors. Preterm Birth: Causes, Consequences, and Prevention. Washington (DC): National Academies Press (US); 2007. Available from http://www.ncbi.nlm.nih.gov/books/NBK11362/ PMID 20669423
- [Background] Garfield CF, Lee Y, Kim HN. Paternal and maternal concerns for their very low-birth-weight infants transitioning from the NICU to home. J Perinat Neonatal Nurs. 2014 Oct-Dec;28(4):305-12. doi: 10.1097/JPN.0000000000000021. PMID 24927295
- [Background] Obeidat HM, Bond EA, Callister LC. The parental experience of having an infant in the newborn intensive care unit. J Perinat Educ. 2009 Summer;18(3):23-9. doi: 10.1624/105812409X461199. PMID 20514124
- [Background] De Rouck S, Leys M. Information needs of parents of children admitted to a neonatal intensive care unit: a review of the literature (1990-2008). Patient Educ Couns. 2009 Aug;76(2):159-73. doi: 10.1016/j.pec.2009.01.014. Epub 2009 Mar 24. PMID 19321288
- [Background] Strauss, A.L., et al., Social organization of medical work. 2nd ed. 1997, New Brunswick, London: Transaction Publishers.
- [Background] Glaser, B.G. and A.L. Strauss, Time for dying. 1968, Chicago, U.S.A.: Aldine
- [Background] Ward K. Perceived needs of parents of critically ill infants in a neonatal intensive care unit (NICU). Pediatr Nurs. 2001 May-Jun;27(3):281-6. PMID 12964668
- [Background] Heermann JA, Wilson ME, Wilhelm PA. Mothers in the NICU: outsider to partner. Pediatr Nurs. 2005 May-Jun;31(3):176-81, 200. PMID 16060580
- [Background] Dhillon AS, Albersheim SG, Alsaad S, Pargass NS, Zupancic JA. Internet use and perceptions of information reliability by parents in a neonatal intensive care unit. J Perinatol. 2003 Jul-Aug;23(5):420-4. doi: 10.1038/sj.jp.7210945. PMID 12847540
- [Background] Kowalski WJ, Leef KH, Mackley A, Spear ML, Paul DA. Communicating with parents of premature infants: who is the informant? J Perinatol. 2006 Jan 1;26(1):44-8. doi: 10.1038/sj.jp.7211409. PMID 16292336
- [Derived] Garfield CF, Kerrigan E, Christie R, Jackson KL, Lee YS. A Mobile Health Intervention to Support Parenting Self-Efficacy in the Neonatal Intensive Care Unit from Admission to Home. J Pediatr. 2022 May;244:92-100. doi: 10.1016/j.jpeds.2022.01.004. Epub 2022 Jan 13. PMID 35033562
- [Derived] Garfield CF, Lee YS, Warner-Shifflett L, Christie R, Jackson KL, Miller E. Maternal and Paternal Depression Symptoms During NICU Stay and Transition Home. Pediatrics. 2021 Aug;148(2):e2020042747. doi: 10.1542/peds.2020-042747. Epub 2021 Jun 18. PMID 34341101